CLINICAL TRIAL: NCT05645926
Title: Association of Obesity and Cardiovascular Outcomes in Patients With Myocardial Infarction : a Korean Nationwide Cohort Study
Brief Title: Association of Obesity and Cardiovascular Outcomes in Myocardial Infarction
Acronym: Paradox
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Kwang-No Lee, Professor, Ajou University School of Medicine
Other Study IDs: AJOUIRB-EXP-2021-398-2
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Obesity Associated Disorder; Myocardial Infarction
Keywords: Obesity paradox; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with MI who underwent revascularization during study period: Patients newly diagnosed with MI and underwent revascularization (PCI or CABG) during study period
  Interventions: Procedure: Percutaneous coronary intervention (PCI); Procedure: Coronary artery bypass grafting (CABG)

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Patients who underwent percutaneous coronary intervention (PCI), including percutaneous transluminal coronary angioplasty (PTCA), and coronary stent insertion
  Other Names: Coronary intervention therapy
Procedure: Coronary artery bypass grafting (CABG) — Patients who underwent coronary artery bypass grafting (CABG)
  Other Names: Coronary graft surgery

SUMMARY:
In this study, the investigators evaluated the association between various measures of adiposity [BMI and waist circumference (WC)] and clinical outcomes in Asian patients with Myocardial Infarction who underwent percutaneous coronary intervention or bypass surgery, using a nationwide population based cohort.

DETAILED DESCRIPTION:
This retrospective nationwide cohort study used administrative claims data from the Korean National Health Insurance Service (NHIS) and the combined health check-up database of the National Health Insurance Corporation between 2013 and 2020.

The investigators included patients newly diagnosed with MI and underwent revascularization (PCI or CABG) between January 2015 and December 2020. Patients aged <20 years, those who were already diagnosed with MI before 2015, and those with cancer were excluded from the analysis. The follow-up period was defined as the time from the index date (date of diagnosis) to each outcome event, date of death, or end of the study period (December 31, 2020), whichever came first.

Patients' demographic data, comorbidities, concomitant medications, and income level were collected from the Korean NHIS database. The recent health check-up data from the index date was also ascertained, including height, weight, waist circumference, blood pressure, health surveys, and laboratory exam. Health survey included family history, smoking history, alcohol history, and the level of individual physical activity.

According to BMI following the World Health Organization recommendation for Asian population, study patients were categorized into 5 groups: underweight, <18.5 kg/m2; normal range, 18.5 to <23 kg/m2; overweight, 23 to <25 kg/m2; obese I, 25 to <30 kg/m2; and obese II, ≥30 kg/m2[4]. The investigators defined the proportion of medical use by calculating formula with the recuperation cost and the number of the visit to hospitals.

During the follow-up period, The investigators assessed 3 clinical outcomes, including all-cause death, cardiovascular hospitalization and the recurrence rate. Clinical outcomes were mainly defined by the the International Classification of Diseases, 10th revision (ICD-10). Patients were censored at the clinical outcomes or the end of the study period (December 31, 2020), whichever came first.

All categorical variables are presented as frequencies and percentages. Normally distributed data were presented as mean ± standard deviation, whereas nonparametric data are presented as median and interquartile range by BMI.

Cox proportional hazard regression analyses were performed to identify the association of BMI with the primary and secondary outcomes, calculating hazard ratio (HR) and 95% confidence interval (CI) and adjusting for the following potential confounders: sex, age, systolic blood pressure, fasting glucose level, total cholesterol level, alcohol consumption, smoking status, physical activity, household income, use of antihypertensive agents, use of statins, use of antiplatelet agents, previous history of MI, previous history of stroke, and index year. All analyses were conducted using R-statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with MI and underwent revascularization (PCI or CABG) between January 2015 and December 2020.

Exclusion Criteria:

* Patients aged <20 years
* Patients diagnosed with MI before 2015
* Patients with cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included patients newly diagnosed with MI and underwent revascularization (PCI or CABG) between January 2015 and December 2020. Patients aged <20 years, those who were already diagnosed with MI before 2015, and those with cancer were excluded from the analysis. The follow-up period was defined as the time from the index date (date of diagnosis) to each outcome event, date of death, or end of the study period (December 31, 2020), whichever came first.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 5 years
  Thromboembolism + Death + CV hospitalization

SECONDARY OUTCOMES:
Thromboembolism | 5 years
  Recurrent myocardial infarction, Stroke
Death | 5 years
  Mortality
CV hospitalization | 5 years
  Admission caused by Cardiovacular disease

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-No LEE, Study Chair — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park SJ, Ha KH, Kim DJ. Body mass index and cardiovascular outcomes in patients with acute coronary syndrome by diabetes status: the obesity paradox in a Korean national cohort study. Cardiovasc Diabetol. 2020 Nov 10;19(1):191. doi: 10.1186/s12933-020-01170-w. PMID 33172464
- [Background] Kim MS, Kim WJ, Khera AV, Kim JY, Yon DK, Lee SW, Shin JI, Won HH. Association between adiposity and cardiovascular outcomes: an umbrella review and meta-analysis of observational and Mendelian randomization studies. Eur Heart J. 2021 Sep 7;42(34):3388-3403. doi: 10.1093/eurheartj/ehab454. PMID 34333589
- [Background] Biswas S, Andrianopoulos N, Dinh D, Duffy SJ, Lefkovits J, Brennan A, Noaman S, Ajani A, Clark DJ, Freeman M, Oqueli E, Hiew C, Reid CM, Stub D, Chan W. Association of Body Mass Index and Extreme Obesity With Long-Term Outcomes Following Percutaneous Coronary Intervention. J Am Heart Assoc. 2019 Nov 5;8(21):e012860. doi: 10.1161/JAHA.119.012860. Epub 2019 Oct 25. PMID 31648578